CLINICAL TRIAL: NCT05637632
Title: Assesslebt of Recombinant HAT-RDT Specificity
Brief Title: Assessment of Recombinant HAT-RDT Specificity
Status: Completed | Type: Observational
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Responsible Party: Sponsor
Other Study IDs: HAT-RDT
Record Dates: First submitted 2022-11-24; First posted 2022-12-05 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Human African Trypanosomiasis
Keywords: rapid diagnostic test; serologic and molecular diagnosis of HAT; neglected tropical disease
MeSH Terms: conditions — Neglected Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample that contains DNA of the Trypanosoma brucei gambiense parasite. the study team will analyse the parasite DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Human African trypanosomiasis HAT, or sleeping sickness, is a tropical disease caused mainly by the parasite Trypanosoma brucei gambiense (gHAT). After a severe epidemic in the 1990s, the World Health Organization (WHO) now targets elimination of transmission of gHAT by the year 2030, which heavily relies on its diagnosis and treatment. Traditional screening tests (like CATT or rapid diagnostic tests (RDTs)) are based on the detection of antibodies against the parasite using native antigens, which are costly and dangerous to produce. New serological tests, using recombinant antigens, have been developed, but little is known about their field performance. The primary objective of this study is to assess the specificity of the newly-developed recombinant RDTs, since it will become very relevant as we move forward towards a screen&treat strategy. We will also compare the diagnostic accuracy and overall performance of iELISA and molecular testing.

DETAILED DESCRIPTION:
This prospective study will follow two different mobile units as they go on their routine screening of the gHAT endemic population. Study participants will be enrolled during the routine screening, and after providing informed consent, they will be asked for a 4.5 ml venous blood sample. The three RDTs (HAT Sero-K-SeT, rHAT Sero-K-SeT, Bioline HAT 2.0) and CATT will be performed on site, while part of the sample will be mixed with DNA/RNA Shield for molecular analysis and the rest will be left to decant, to collect plasma for iELISA and TL. Confirmatory tests will be performed in the field on any seropositive individual. Should any case be confirmed, treatment will be offered, free of charge, following PNLTHA guidelines.

The obtained data will allow for a very precise estimation of the specificity of the newly developed recombinant RDTs. This study does not aim to determine the sensitivity of these tests since, due to the very low prevalence, the chance of having sufficient seropositive samples and/or finding a true case are very slim. The diagnostic performance of iELISA and novel molecular tests will also be determined.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent (and assent for minors 12-17years old)
* Be enrolled in routine HAT screening activities dony by the mobile unit (PNLTHA mobile unit routine active screening teams that visit villages at risk for HAT). People living in the village are targeted for screening.
* Participants must be at least 12 years old

Exclusion Criteria:

* Chilrden younger than 12 years old
* previously treated for HAT
* refusal to provide informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population are the people living in villages that are at risk for HAT infection, as the first stade of the disease is asymptomatic or with non-specific symptoms, the whole village is invited to participate in the active screening activity. This is routine active screening done by the mobile team. they study team will recruit people that participate to the screening campaign.
Sampling Method: Non-Probability Sample
Enrollment: 1504 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Specificity of recombinant CORIS rapid diagnostic test for HAT | 1 month
  recombinant RDT for detection of HAT developed by CORIS, determine its field performance
Specificity of recombinant BIOLINE rapid diagnostic test for HAT | 1 months
  recombinant RDT for detection of HAT developed by BIOLINE, determine its field performance

SECONDARY OUTCOMES:
iELISA | 3 months
  determine performance of inhibition ELISA test to replace Trypanolyse test
Molecular | 4 months
  determine if active infection of HAT is present using molecular testing technique, determine its performances

CONTACTS AND LOCATIONS:
Overall Officials: Epco Hasker, Phd PH, Study Director — Insitute of Tropical Medicine
Locations (1):
- Programme National de Lutte contre la Trypanosomiase Humaine Africaine (PNLTHA), Kinshasa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: Undecided
anonymity of participants must be guaranteed anonymised study results can be shared with other researchers

REFERENCES:
- [Derived] Tablado Alonso S, Inocencio Da Luz R, Van Reet N, Ngay I, Pemba MM, Roge S, Kwete J, Nicco E, Rigouts L, Miaka EM, Ngoyi DM, Verle P, Buscher P, Hasker E. Prospective evaluation of 2nd generation rapid diagnostic tests for the serological diagnosis of gambiense human African trypanosomiasis in the Democratic Republic of the Congo. BMC Infect Dis. 2025 Dec 6;26(1):46. doi: 10.1186/s12879-025-12278-3. PMID 41351066